CLINICAL TRIAL: NCT02121925
Title: LUNG CAncerREgistry: An Open Registry to Measure the Impact of Adding RNA Expression Testing (myPlan Lung Cancer) on Referral Decisions and to Assess Disease-free Survival With Long-term Follow-up in Newly Diagnosed Early Stage Lung Adenocarcinoma Patients
Brief Title: Registry Measuring the Impact of Adding RNA Expression Testing on Referral Decisions in Early Stage Lung Cancer Patients and Assessing the Disease-free Survival With Long-term Follow-up
Acronym: ONC003
Status: Terminated | Type: Observational
Why Stopped: Company decision to terminate
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: myPlan ONC003
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2015-09

CONDITIONS: Lung Cancer; NSCLC; Lung Adenocarcinoma
Keywords: Registry
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tissue from blocks or slides of prostatic adenocarcinoma biopsies.
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry is intended to measure the effect of myPlan Lung Cancer™ test has on treatment decisions of Surgeons when added to standard clinical-pathological parameters in patients with early stage NSCLC.The sponsor is conducting two parallel registries, with one directed at Surgeons (ONC003) and the other at Oncologists (ONC006).This registry is specific to Surgeons (ONC003). Outcomes measures on lung cancer relapse and death from any cause will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage non-small cell lung adenocarcinoma
* Sub-population staging (IA, IB or IIA) as judged by the standard of practice at the investigational site
* Resection of tumor within previous 2 months of enrollment
* ECOG performance of 0-2
* A minimum life expectancy of six months

Exclusion Criteria:

* Pre-operative radiation or chemotherapy for NSCLC
* Post-operative radiation or chemotherapy for NSCLC
* Enrollment in a separate clinical trial restricting treatment options
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed treatment-naïve patients with early stage NSCLC (lung adenocarcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2014-05; Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage change from Pre-Test to Post-Test referral | 3 months
  The percentage change from the recorded PRE-TEST referral by surgeon versus the POST-TEST referral following results of myPlan Lung Cancer testing

SECONDARY OUTCOMES:
Percentage change from the Pre-test referral to the 60-day Post-Test referral | 2 months
  The percentage change from the recorded Pre-Test referral by surgeon versus the 60 day post-test actual referral attendance
Percentage of patients at 60 days post test receiving treatment | 2 months
  The percentage of patients at 60 day post-test who are receiving radiation and or chemotherapy treatment
Percentage change from Pre-Test to Post-Test chest surveillance plan | 3 months
  The percentage change from the recorded Pre-Test chest surveillance plan versus the Post-Test chest surveillance plan
Assessment of disease free survival from resection to relapse or death | 3 years
  Disease-free survival, which is defined as the time from resection to the first of two events: lung cancer relapse or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (1):
- Seattle, Washington, United States